CLINICAL TRIAL: NCT02020122
Title: Pain Prevention and Treatment Through the Enhancement of the Anti-nociceptive Component of Pain Modulation Profiles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, d_yarnitsky, Professor, Head of Neurology Deapartment, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0472-13-RMB.CTIL
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Pain
Keywords: endogenous pain modulation; coronary artery bypass grafting; quantitative sensory testings; duloxetine; pregabalin; preemptive treatment
MeSH Terms: conditions — Pain | interventions — Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Duloxetine (Active Comparator): DUL 60mg x once a day x 2 days. This arm will also take 2 non-active placebo x once a day x 2 days
  Interventions: Drug: Duloxetine; Drug: Placebo
- Pregabalin (Active Comparator): PGB 150mg x twice a day x 2 days
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Non active placebo x twice a day x 2 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — duloxetine 60mg
  Arms: Duloxetine
Drug: Pregabalin — pregabalin 150mg
  Arms: Pregabalin
Drug: Placebo — non active placebo
  Arms: Duloxetine; Placebo

SUMMARY:
To utilize the plasticity of the central pain pathways in order to (i) shift individuals with a pro-nociceptive pain modulation profile towards an anti-nociceptive one, and (ii) assess its relevance in minimizing pain-derived morbidity.

DETAILED DESCRIPTION:
In the project proposed here our main aim is to shift pain modulation towards anti-nociception as a novel approach to pain prevention and treatment. Our first hypothesis is that individual's modulation profile, when not anti-nociceptive, can be pharmacologically shifted into being anti-nociceptive. We assert (the first hypothesis) that such shift can be optimized by coupling the drug's mode of action with the individual's pain modulation profile; based on limited available data, it is suggested that less efficient inhibitory pain modulation will be modified best by serotonin-norepinephrine reuptake inhibitors (SNRIs), whereas enhanced facilitatory modulation will be modified best by Ca++ channel ligands. Pain modulation will be assessed by psychophysical tools, and will include dynamic tests of pain modulation. The conditioned pain modulation (CPM) test protocol will be used for assessing pain inhibition, and the temporal summation (TS) test protocol will be used for assessment of pain facilitation. Our second hypothesis is that SNRIs will be most efficacious in shifting individuals into being antinociceptive if these individuals had lower activation of the anterior brain pain network in the CPM test paradigm. In turn, Ca++ channel ligands will be most efficacious for individuals showing enhanced activation of the posterior pain network sites in response to the TS test protocol. Our third hypothesis is that an anti-nociceptive pain modulation profile protects individuals from acquiring pain. The model we chose for this study is surgery for coronary artery bypass grafting (CABG). Individuals scheduled for surgery, who are pain free, will be assigned to 3 arms - (1) duloxetine (DUL) (SNRI), (2) pregabalin (PGB) (Ca++ channel ligand) and (3) placebo. Drugs will be taken for 48 hours prior to surgery in a double-blind non cross-over parallel design. Pain modulation will be assessed before treatment, 2-4 hours prior to surgery and at its end, 6 weeks before surgery. Post operative acute and chronic pain will be assessed up to 2 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy, age 18-75.

Exclusion Criteria:

* Regular use of analgesia for any purpose, including SNRIs, gabapentins, COX inhibitors.
* Presence of diagnosed chronic pain disorders, psychiatric disorders, cognitive and /or neurological deficit.
* Inability to give informed consent, communicate and understand the purpose and instructions of this study.
* Pregnant or nursing women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The changes in pain response after administration of duloxetine and pregabalin | 3 years
  The changes in the excitatory and inhibitory pain modulation responses (assessed by temporal summation and conditioned pain modulation) will be examined before and after the administration of duloxetine and pregabalin in the set of pre and post coronary artery bypass grafting surgery.

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, Professor, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel